CLINICAL TRIAL: NCT01865565
Title: A Trial for Surgical Treatment in Patients With Initially Locally Unresectable Advanced GIST Without Metastasis During Therapy With Imatinib
Brief Title: Surgery for Locally Unresectable Advanced GISTs Without Metastasis After Imatinib Therapy
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chun-Nan Yeh, MD, Associate Professor, Dept. of General Surgery., Chang Gung Memorial Hospital
Other Study IDs: Yeh CN001
Record Dates: First submitted 2013-05-22; First posted 2013-05-31 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: gastrointestinal stromal tumor; GIST; neoadjuvant; imatinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Histologically verified GIST and exon genotype.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Imatinib treat: • Locally advanced unresectable GIST without metastasis at
  * EC junction requiring total gastrectomy,
  * Duodenum requiring Whipple operation;
  * Large GIST requiring multiviceral resection;
  * Rectum: requiring APR.

SUMMARY:
Gastrointestinal stromal tumors (GISTs) are a form of sarcoma and the most common sarcoma tumors of the gastrointestinal tract. The limited clinical experience suggests that GIST patients may benefit from neo-adjuvant therapy from primary GIST. This is a prospective, multicenter, open, observational study in evaluation of safety and efficacy of imatinib compared with that of historical data for locally unresectable advanced GIST without metastasis. The study will include an up to 28-day screening period, followed by receiving imatinib mesylate (400 mg/day) for at least 6-12 months and followed up for 3 years after surgery.

DETAILED DESCRIPTION:
Primary Objective

* To observe the safety of imatinib compared with that of historical data for locally unresectable advanced GIST without metastasis.

Secondary Objective

* Progression-free survival (PFS) in resected patients during follow up
* R0 resection rate
* objective response rate, tumor shrinkage rate
* Correlation of mutation status with response
* Correlation of PK with response
* Surgical morbidity and mortality and safety follow up
* Quality of life
* Overall survival (OS)

ELIGIBILITY:
Inclusion Criteria

* Locally advanced unresectable GIST without metastasis at

  * EC junction requiring total gastrectomy,
  * Duodenum requiring Whipple operation;
  * Large GIST requiring multiviceral resection;
  * Rectum: requiring APR.
* Histologically documentation with positive immunostaining for KIT (CD117)
* Patient age ≥ 18 years old
* ECOG performance status 0 or 1
* Patient must have the following post-operative laboratory values confirmed within 14 days prior to registration:

  * Creatinine ≤ 1.5 times the institution ULN (upper limit of normal)
  * WBC ≥ 3,000/mm3
  * Platelets ≥ 100,000/mm3
  * Total Bilirubin ≤ 1.5 times the institution ULN. NOTE: Patients with elevated bilirubin secondary to Gilbert's disease are eligible to participate in the study.
  * AST ≤ 2.5 times the institution ULN
  * ALT ≤ 2.5 times the institution ULN
  * Female of childbearing potential must have negative serum pregnancy test. -- -NOTE: Post-menopausal women must be amenorrheic for at least 12 months to be deemed not of reproductive potential.
* Patient is willing to sign informed consent.

Exclusion Criteria

* Patient has received post-operative chemotherapy.
* Patient has received post-operative radiation therapy.
* Patient has received post-operative investigational treatment.
* Patient has received prior therapy with imatinib, or any other molecular targeted or biological therapy.
* Patient has had an active infection requiring antibiotics within 14 days prior to registration.
* any prior malignancies for at least 5 years with potential evidence of recurrence (except for effectively treated basal cell or squamous carcinoma of the skin, carcinoma in-situ of the cervix that has been effectively treated by surgery alone, or lobular carcinoma in-situ of the ipsilateral or contralateral breast treated by surgery alone).
* Patient is deemed by their treating physician to be at risk for recurrence from prior malignancies.New York Heart Association Class 3 or 4 cardiac diseases.
* Patient is taking full dose warfarin. NOTE: The use of mini-dose warfarin (1 mg orally per day) for prevention of central line-associated deep venous thrombosis is permitted.
* Presence of severe and/or uncontrolled concurrent medical disease (e.g., uncontrolled diabetes, uncontrolled chronic renal disease, uncontrolled liver disease, including chronic viral hepatitis judged at risk of reactivation, uncontrolled active infection, such as HIV infection, etc.).
* Patient, if female and breastfeeding. NOTE: It is not known whether imatinib or its metabolites are excreted in human milk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in four branch hospitals of Chang Gung Memorial Hospital, Taiwan including Keelung, Linkou, Cha-Yi, and Kaoshung, respectively. To target 50 patients; 90% patients with response after imatinib treatment; 10% patients without response; compare the result with historical data.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
progression free survival | five years
  Evidence of measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines with CT scan.

SECONDARY OUTCOMES:
R0 resection rate | three years
  all the participants
Objective response rate, tumor shrinkage rate | three years
  all the participants
Correlation of PK with response | three years
  check PK (trough level of imatinib)of all the participants at first month and every three months later to correlate with the response and check PK (peak level of imatinib) of all the participants who had adverse events
Surgical morbidity and mortality and safety follow up | five years
  surgical morbidity: morbidity related to surgical procedure surgical mortality: mortality related to surgical procedure safety: adverse events related imatinib according to NIH toxicity evaluation criteria
Overall survival (OS) | five years
  Overall survival (OS) will be measured from after administration of imatinib mesylate and death as the end point of the study, whatever the cause. Alive patients will be censored at the date of last follow-up. Causes of death will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Nan Yeh, MD, Study Chair — Chang Gung Memorial Hospital, Linkou, Taiwan.; Jen-Shi Chen, MD., Principal Investigator — Chang Gung Memorial Hospital, Linkou, Taiwan.; Yen-Yang Chen, MD., Principal Investigator — Chang Gung Memorial Hospital, Kaoshung, Taiwan.; Kun-Chun Chiang, MD., Principal Investigator — Chang Gung Memorial Hospital, Keelung, Taiwan.; Liang-Mou Kuo, MD., Principal Investigator — Chang Gung Memorial Hospital, Cha-Yi, Taiwan.
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Background] Pawlik TM, Vauthey JN, Abdalla EK, Pollock RE, Ellis LM, Curley SA. Results of a single-center experience with resection and ablation for sarcoma metastatic to the liver. Arch Surg. 2006 Jun;141(6):537-43; discussion 543-4. doi: 10.1001/archsurg.141.6.537. PMID 16785353
- [Background] Dagher R, Cohen M, Williams G, Rothmann M, Gobburu J, Robbie G, Rahman A, Chen G, Staten A, Griebel D, Pazdur R. Approval summary: imatinib mesylate in the treatment of metastatic and/or unresectable malignant gastrointestinal stromal tumors. Clin Cancer Res. 2002 Oct;8(10):3034-8. PMID 12374669
- [Background] Demetri GD, von Mehren M, Blanke CD, Van den Abbeele AD, Eisenberg B, Roberts PJ, Heinrich MC, Tuveson DA, Singer S, Janicek M, Fletcher JA, Silverman SG, Silberman SL, Capdeville R, Kiese B, Peng B, Dimitrijevic S, Druker BJ, Corless C, Fletcher CD, Joensuu H. Efficacy and safety of imatinib mesylate in advanced gastrointestinal stromal tumors. N Engl J Med. 2002 Aug 15;347(7):472-80. doi: 10.1056/NEJMoa020461. PMID 12181401
- [Background] Blanke CD, Rankin C, Demetri GD, Ryan CW, von Mehren M, Benjamin RS, Raymond AK, Bramwell VH, Baker LH, Maki RG, Tanaka M, Hecht JR, Heinrich MC, Fletcher CD, Crowley JJ, Borden EC. Phase III randomized, intergroup trial assessing imatinib mesylate at two dose levels in patients with unresectable or metastatic gastrointestinal stromal tumors expressing the kit receptor tyrosine kinase: S0033. J Clin Oncol. 2008 Feb 1;26(4):626-32. doi: 10.1200/JCO.2007.13.4452. PMID 18235122